CLINICAL TRIAL: NCT04107740
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IV Clinical Trial to Evaluate and Compare the Efficacy and Safety of C-Trelin OD Tab 5mg(Taltirelin Hydrate) in Patients With Ataxia Induced by Spinocerebellar Degeneration
Brief Title: C-Trelin Orally Disintegrated(OD) Tablet 5mg in Ataxia Due to Spinocerebellar Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HLB Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTT-004
Record Dates: First submitted 2019-09-10; First posted 2019-09-27 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-02

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration; Ataxia
MeSH Terms: conditions — Spinocerebellar Degenerations; Ataxia | interventions — TA 0910

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-Trelin OD Tab(5mg Taltirelin Hydrate) (Experimental): BID, 10mg per day, for 24 weeks
  Interventions: Drug: C-Trelin OD Tab(5mg Taltirelin Hydrate)
- Placebo (0mg Taltirelin Hydrate) (Placebo Comparator): BID, 10mg per day, for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C-Trelin OD Tab(5mg Taltirelin Hydrate) — BID, 10mg per day, for 24 weeks
  Arms: C-Trelin OD Tab(5mg Taltirelin Hydrate)
Drug: Placebo — BID, 10mg per day, for 24 weeks
  Arms: Placebo (0mg Taltirelin Hydrate)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of C-Trelin OD Tablet 5mg(Taltirelin Hydrate) in Multicenter, randomized, double-blind, placebo-controlled clinical trial in patients with ataxia induced by spinocerebellar degeneration.

DETAILED DESCRIPTION:
Taltirelin Hydrate, an active substance of C-Trelin OD tablet 5mg, is an analogue of Thyrotropin Releasing Hormone(TRH). TRH is distributed widely in the brain, and exerts variety of central nervous system effects as well as endocrine activity such as releasing of Thyroid Stimulating Hormone(TSH) and Prolactin. Based on these actions, studies have been attempted for the treatment of various neurological diseases such as refractory epilepsy, cerebellar ataxia, amyotrophic lateral sclerosis, cerebellar ataxia and so on. C-Trelin OD tablet 5mg(Taltirelin Hydrate), an investigational product, is a commercially available drug that was approved by Ministry of Food and Drug Safety(MFDS) based on the safety and efficacy. However, the studies with this medicine were conducted before 1997, and the evaluation criteria for the efficacy was quite different from the current evaluation criteria.

In this clinical trial, K-SARA as an objective evaluation criteria validated in Korean patients is used to confirm the efficacy of C-Trelin to improve ataxia, and to prove safety by evaluating changes in clinical laboratory data and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 20 years of age
* Patients who voluntarily agreed to enroll in the study and signed an informed consent form
* Patients diagnosed with ataxia (genetic or non-genetic) due to spinocerebellar degeneration by the investigator's judgment based on the results of essential diagnostic examinations stated below.

<Genetic ataxia>

* Spinocerebellar ataxia(SCA)
* Friedreich's ataxia(FA)
* Other genetic ataxia

<Non-genetic ataxia>

* Idiopathic late onset cerebellar ataxia(ILOCA) The following examinations to diagnose ataxia (genetic or non-genetic) induced by spinocerebellar degeneration can be used, and the investigator has to diagnose by combining at least one diagnostic examination result among the following-items.
* Medical history: alcohol abuse, medication history, family history
* Genetic test: SCA 1, 2, 3, 6, 7, 8, 17, FA which is available for the patient
* Brain MRI or CT scan: abnormalities of cerebellum and pons, brain vascular disease, or brain tumors
* Retinal or optic nerve examination

Exclusion Criteria:

* Patients with bed-ridden state at the time of screening even though the patient is diagnosed with ataxia induced by spinocerebellar degeneration
* Patients with ataxia caused by stroke
* Patients with ataxia caused by cerebrovascular, alcoholic-induced or drug-induced secondary cerebellar abnormalities
* Patients with complications of other neurodegenerative diseases such as Parkinson's disease and multiple system atrophy(however, patients diagnosed with SCA 2, SCA 3, SCA 17 can be enrolled)
* Patients with malignant neoplastic disease
* Patients with kidney failure and liver failure history
* Patients with abnormalities in clinical laboratory test results as follows( Patients with liver dysfunction: Aspartate Transaminase(AST), Alanine Transaminase(ALT) > 3 times than the upper limit of normal range(ULN), Total bilirubin > 1.5 times than the ULN, Patients with renal dysfunction: Serum creatinine > 1.5mg/dl, Patients with thyroid dysfunction: free T4: above or below the normal range)
* Patients with thyroid dysfunction at the time of screening(hyperthyroidism, hypothyroidism)
* Patients accompanied by lesions other than spinocerebellar degeneration from Brain MRI or CT scan
* Patients with schizophrenia, major depressive disorder
* Patients with a history of acute myocardial infarction within 2 years of the screening visit
* Patients with a history of unstable angina pectoris within 2 years of the screening visit
* Patients taking contraindicated concomitant medication( However, patients with following drugs can be enrolled only if they are administered 4 weeks before the screening visit, and the type, dosage, and volume should be kept unchanged during the clinical trial.: Parkinson's disease medicine, Anxiolytics, Antidepressants, Antiepileptics, Antipsychotics, Medicine for dysuria, Sleep inducer, β blocker)
* Patients with hypersensitivity to Taltirelin Hydrate
* Cognitive dysfunction: Korean Version of Mini-Mental State Exam(K-MMSE) ≤ 20
* Patients who are pregnant or lactating
* All childbearing females who are planning to pregnant during the clinical trial or who are not using medically reliable contraceptive methods (such as intrauterine contraceptives, condoms or diaphragms combined with spermicides) except menopaused more than 1 year from the last menstruation or had undergone surgical sterilization
* Patients participating in any other clinical trials or participated 30 days before
* Patients whom the investigator considers inappropriate for the clinical trial due to any other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Changes in Korean Version of Scale for the Assessment and Rating of Ataxia(K-SARA) scores | 24 weeks of administration compared to the baseline
  K-SARA consists of walking, standing, sitting, speech impairment, finger following, nose-finger test, palm flipping, and heel-shin test. The total score is 40 and higher scores indicate serious ataxia.

SECONDARY OUTCOMES:
Changes in Korean Version of Scale for the Assessment and Rating of Ataxia(K-SARA) scores | 4 weeks and 12 weeks of administration compared to the baseline
  K-SARA consists of walking, standing, sitting, speech impairment, finger following, nose-finger test, palm flipping, and heel-shin test. The total score is 40 and higher scores indicate serious ataxia.
Changes in Clinical Global Impression - Severity(CGI-S) scores | 4 weeks, 12 weeks, and 24 weeks of administration compared to the baseline
  Changes in Clinical Global Impression(CGI) is a commonly used measure to assess the severity of symptoms, improvement, the effectiveness of treatment and it consists of Clinical Global Impression-Severity(CGI-S), Clinical Global Impression-Improvement scale(CGI-I), and Clinical Global Impression-Efficacy index(CGI-E). Clinical Global Impression-Severity(CGI-S) means overall clinical impression at the time of drug administration. It ranges from 1 to 7, higher scores indicate higher severity.
Changes in Clinical Global Impression - Improvement(CGI-I) scores | 12 weeks and 24 weeks of administration compared to 4 weeks of administration
  Changes in Clinical Global Impression(CGI) is a commonly used measure to assess the severity of symptoms, improvement, the effectiveness of treatment and it consists of Clinical Global Impression-Severity(CGI-S), Clinical Global Impression-Improvement scale(CGI-I), and Clinical Global Impression-Efficacy index(CGI-E). Clinical Global Impression-Improvement scale(CGI-I) means current improvement from the patient's baseline status. It ranges from 1 to 7, and higher scores indicate worsening of symptoms.
Changes in Clinical Global Impression - Efficacy index(CGI-E) scores | 12 weeks and, 24 weeks of administration compared to 4 weeks of administration
  Changes in Clinical Global Impression(CGI) is a commonly used measure to assess the severity of symptoms, improvement, the effectiveness of treatment and it consists of Clinical Global Impression-Severity(CGI-S), Clinical Global Impression-Improvement scale(CGI-I), and Clinical Global Impression-Efficacy index(CGI-E). Clinical Global Impression-Efficacy index(CGI-E) indicates the effect of the current treatment and the severity of the side effects. It is calculated by dividing the treatment effect by the side effects. The treatment effect ranges from 1 to 4, and higher scores indicate the better effect. The side effect ranges from 1 to 4, and higher scores indicate the greater side effect.
Changes in Korean Version of the Scale for Outcomes in Parkinson's Disease-Autonomic(K-SCOPA-AUT) scores | 24 weeks of administration compared to the baseline
  Korean Version of the Scale for Outcomes in Parkinson's Disease-Autonomic(K-SCOPA-AUT) score is a patient report questionnaire for intensive evaluation of autonomic dysfunction in Parkinson's disease to determine the problems with physical functioning, such as difficulty in urinating or sweating over the past month. The total score is 69 points, and each item is evaluated on a scale of 0(never) to 3(often).
Changes in EQ-5D-5L scores | 24 weeks of administration compared to the baseline
  EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ Visual Analogue Scale (EQ VAS). EQ-5D-5L descriptive system consists of 5 items (mobility, self-care, usual activities, pain / discomfort, anxiety / depression), and 5 levels for each item [No problems (Level 1), slight problems (Level 2), moderate problems (Level 3), severe problems (Level 4), extreme problems (Level 5)]. EQ Visual Analogue Scale(EQ VAS) measures and records the subject's rating for their current health-related quality of life state on a 20cm visual analogue scale. Each endpoint is marked with "best imaginable health(100)" and "worst imaginable health(0)".
Changes in Tinetti balance test & Gait assessment scores | 24 weeks of administration compared to the baseline
  Tinetti balance test & Gait assessment measures the gait and balance of a subject according to the subject's ability to perform a specific task. Each item is scored by 0 to 2 and higher scores indicate the better performance. The sum of each individual score consists of the total gait scores(12 points), the total balance scores(16 points), and the sum of the gait and balance scores(28 points).

CONTACTS AND LOCATIONS:
Overall Officials: Seong-beom Koh, Principal Investigator — Korea University Guro Hospital
Locations (8):
- South Korea (8):
  - Chonnam National University Hospital, Gwangju
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No